CLINICAL TRIAL: NCT02016261
Title: Open Label, Non-comparative Study to Evaluate Cognitive Functioning in Remitted Depression Outpatients During Long-term Preventive Treatment With Fluvoxamine
Brief Title: Study to Evaluate Cognitive Functioning in Remitted Depression During Treatment With Fluvoxamine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Moscow Research Institute of Psychiatry (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A13-996
Record Dates: First submitted 2013-12-10; First posted 2013-12-19 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Recurrent Depressive Disorder
Keywords: Cognitive function
MeSH Terms: conditions — Depressive Disorder | interventions — Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remitted Depression Outpatients (Experimental): Adults 18-65 years old, males and females with the diagnosis of recurrent depressive disorder and who had at least two severe depressive episodes (with or without psychotic symptoms) of the disorder and who currently in remission
  Interventions: Drug: Fluvoxamine

INTERVENTIONS:
Drug: Fluvoxamine — The subjects will be prescribed Fluvoxamine treatment for 24 weeks with dose 50-300 mg
  Other Names: Fevarin®

SUMMARY:
Open label, non-comparative, prospective study to evaluate cognitive functioning in remitted depression outpatients during long-term preventive treatment with Fluvoxamine (Fevarin®)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of recurrent depressive disorder at least two years prior to enrollment into the study.
2. At least two severe depressive episodes with or without psychotic symptoms in the past medical history.
3. Stable patient in remission since at least 4 weeks after depressive episode and not more than 6 months after depressive episode.
4. Planned prescription of fluvoxamine for preventive therapy in recurrent depressive disorder.
5. The subject is fluent in Russian language.
6. According to Stroop test one of following points has to be met - increase of the words reading time on 10% and more or three and more mistakes done.
7. Sum of Addenbrooke's Cognitive Examination total scores must be 93 or less.
8. Male or female, between the ages of 18 and 65 years.
9. If female, postmenopausal or birth control.

Exclusion Criteria:

1. Diagnosis of the following concomitant psychiatric disorders: current depressive or maniac episode, bipolar affective disorder, persistent mood affective disorder (cyclothymia, dysthymia, other or unspecified persistent mood disorder), other or unspecified mood affective disorder, substance-related disorders, schizophrenia, or other psychotic disorders.
2. History of a drug or alcohol disorder.
3. Current treatment with fluvoxamine.
4. History of depressive disorder associated with endocrine disorders.
5. Pregnancy, breast-feeding female patients.
6. History of any significant neurologic disease.
7. Treatment with electroconvulsive therapy in the 6 months preceding the study.
8. Major risk of suicide.
9. Hypersensitivity to fluvoxamine.
10. Use of the medications, which are known to interact with fluvoxamine.
11. Have initiated psychotherapy or other therapies (such as acupuncture or hypnosis).
12. Have initiated cognitive remediation therapy within 12 weeks prior enrollment or at any time during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change of time difference between Part I and Part II of Stroop Test | From baseline up to Week 24

SECONDARY OUTCOMES:
Change of total Frontal Assessment Battery score | From baseline up to Week 24
Proportion of patients maintained remission status | Week 24
Changes of Addenbrooke's Cognitive Examination general score | From baseline up to Week 24
Change of The Social Adaptation Self-evaluation Scale total score | From baseline up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Alexey E. Bobrov, Professor, Principal Investigator — Moscow Research Institution of Psychiatry
Locations (1):
- Moscow Research Institution of Psychiatry, Moscow, Russia